CLINICAL TRIAL: NCT03691545
Title: Helping Rural-living Young Adult Cancer Survivors Make Healthy Lifestyle Choices: Does Having a Telehealth Personal Health Coach Help?
Brief Title: Making Healthy Choices: Does Having an Online Health Coach Help?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Associate Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H08-18-882
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Physical Activity; Dietary Modification
Keywords: physical activity; fruit and vegetable consumption; telehealth; young adult cancer survivors; rural-dwelling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): (1) 12 weekly interactive sessions with a health coach to help them set goals and make changes toward becoming physically active and consuming the recommended number of fruits and vegetables.
  Interventions: Behavioral: interactive sessions

INTERVENTIONS:
Behavioral: interactive sessions — This arm will receive personalized health coaching (behaviour change counseling)

SUMMARY:
Participating in regular physical activity and consuming a diet high in fruits and vegetables can aid in the management of various acute and chronic side effects of cancer treatment; however, few rural-dwelling young adult cancer survivors are active enough and consume enough fruits and vegetables to accrue benefits. Telehealth interventions show promise for helping these young adults increase their motivation to participate in these behaviours by addressing barriers associated with accessing face-to-face behaviour counselling services (e.g., time commitment, travel distance). Yet, few researchers have examined the feasibility and acceptability of a telehealth intervention that provides motivational support grounded in self-determination theory for these health behaviours in rural-dwelling young adult cancer survivors. Based on previous research, the researchers reasoned that rural-dwelling young adult cancer survivors' physical activity and fruit and vegetable consumption would be more likely to increase if they participated in a telehealth intervention therefore, the researchers aim to test the feasibility, acceptability, and preliminary efficacy of the intervention. The researchers also aim to assess if changes in perceived basic psychological need satisfaction, behaviour regulation, and perceived autonomy support are associated with changes in physical activity and fruit and vegetable consumption.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 20-39 years
* Live in a rural area (i.e., areas with <35,000 inhabitants)
* Have completed primary treatment for non-metastatic cancer
* Are not currently meeting the American Cancer Society guidelines for physical activity and fruit and vegetable consumption
* Have access to the Internet and to audio-visual devices
* Are willing to provide informed consent to participate in this study and willing to follow study protocol
* Able to read and understand English
* Are ambulatory

Exclusion Criteria:

* Have a serious condition that precludes safe participation in physical activity
* Have symptomatic heart or vascular diseases (angina, peripheral vascular disease, congestive heart failure)
* Have severe hypertension
* Have had a recent stroke
* Have a chronic obstructive pulmonary disease
* Have severe insulin-dependent diabetes mellitus
* Have renal disease
* Have liver disease

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Physical activity behaviour: International Physical Activity Questionnaire Short Form (IPAQ-S; Booth, 2000). | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported physical activity (over the past 7 days) from baseline to post-intervention, with higher scores representing a better outcome.
Fruit and vegetable intake behaviour: Behavioural Risk Factor Surveillance System Fruit and Vegetable section (BRFSS-FV; Trowbridge, Wong, Byers, & Serdula, 1990) | Baseline (week 0) and post-intervention (week 12)
  Change in self-reported fruit and vegetable intake (over the past 7 days) from baseline to post-intervention, with higher scores representing a better outcome.

SECONDARY OUTCOMES:
Basic psychological needs satisfaction for physical activity: Psychological Need Satisfaction in Exercise Scale (PNSE; Wilson, Rogers, Rodgers, & Wild, 2006) | Baseline (week 0) and post-intervention (week 12)
  Change in basic psychological need satisfaction for physical activity from baseline to post-intervention, using a 1 (false) to 6 (true) scale with higher scores representing a better outcome.
Basic psychological need satisfaction for fruit and vegetable consumption: Psychological Need Satisfaction questionnaire (PNS; Deci, Ryan, Gagne, Leone, Usunov, & Kornazheva, 2001) | Baseline (week 0) and post-intervention (week 12)
  Change in basic psychological need satisfaction for fruit and vegetable consumption from baseline to post-intervention, using a 1 (strongly disagree) to 7 (strongly agree) scale with higher scores representing a better outcome.
Motivational regulations for physical activity: Exercise Treatment Self-Regulation Questionnaire (TSRQ-E; Williams, Deci, & Ryan, 1998) | Baseline (week 0) and post-intervention (week 12)
  Change in motivational regulations for physical activity from baseline to post-intervention, using a 1 (not at all true) to 7 (very true) scale with higher scores representing a better outcome.
Motivational regulations for fruit and vegetable consumption: Dietary Self-Regulation questionnaire (DSR; Williams, Deci, & Ryan, 1998) | Baseline (week 0) and post-intervention (week 12)
  Change in motivational regulations for fruit and vegetable consumption from baseline to post-intervention, using a 1 (not at all true) to 7 (very true) scale with higher scores representing a better outcome.
Perceived autonomy support: Health Care Climate Questionnaire (HCCQ; Williams, Grow, Freedman, Ryan, & Deci, 1996) | Post-intervention (week 12)
  Level of perceived autonomy support for health behaviours post-intervention, using a 1 (strongly disagree) to 7 (strongly agree) scale with higher scores representing a better outcome.
Recruitment rates | Duration of recruitment and intervention phase (12 weeks)
  The number of eligible participants who enrol in the study out of the number assessed for eligibility
Retention rates for intervention | Duration of recruitment and intervention phase (12 weeks)
  The number of participants completing the 12-week intervention.
Adherence rates for intervention | Duration of recruitment and intervention phase (12 weeks)
  The number of eligible participants completing ≥ 70% of the intervention sessions (i.e., 8/12)
Acceptability of intervention: Semi-structured interviews | Post-intervention (12 weeks)
  Participants will be asked what they liked, disliked, and experienced during the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Booth M. Assessment of physical activity: an international perspective. Res Q Exerc Sport. 2000 Jun;71(2 Suppl):S114-20. No abstract available. PMID 10925833
- [Background] Deci, E. L., Ryan, R.M., Gagne, M., Leone, D.R., Usunov, J., & Kornazheva, B.P. (2001). Need satisfaction, motivation, and well-being in the work organizations of a former eastern bloc country: A cross-sectional study of self-determination. Journal of Personality and Social Psychology, 27(8), 930-942.
- [Background] Trowbridge FL, Wong FL, Byers TE, Serdula MK. Methodological issues in nutrition surveillance: the CDC experience. J Nutr. 1990 Nov;120 Suppl 11:1512-8. doi: 10.1093/jn/120.suppl_11.1512. PMID 2173743
- [Background] Williams, G. C., Deci, E. L., & Ryan, R. M. (1998). Building health-care partnerships by supporting autonomy: Promoting maintained behavior change and positive health outcomes. In A. L. Suchman, P. Hinton-Walker, & R. Botelho (Ed.), Partnerships in healthcare: Transforming relational process (pp. 67-87). Rochester, NY: University of Rochester Press.
- [Background] Williams GC, Grow VM, Freedman ZR, Ryan RM, Deci EL. Motivational predictors of weight loss and weight-loss maintenance. J Pers Soc Psychol. 1996 Jan;70(1):115-26. doi: 10.1037//0022-3514.70.1.115. PMID 8558405
- [Background] Wilson, P. M., Rogers, W. T., Rodgers, W. M., & Wild, T. C. (2006). Psychological need satisfaction in exercise scale. Journal of Sport & Exercise Psychology, 28, 231-251.
- [Derived] Price J, Brunet J. Feasibility and acceptability of a telehealth behavior change intervention for promoting physical activity and fruit and vegetable consumption among rural-living young adult cancer survivors. J Psychosoc Oncol. 2021;39(6):715-733. doi: 10.1080/07347332.2021.1896616. Epub 2021 Apr 2. PMID 33798033